CLINICAL TRIAL: NCT07400991
Title: Restrictive Versus Liberal Fluid Intake in Acute Decompensated Heart Failure: a Randomized Trial
Brief Title: Restrictive Versus Liberal Fluid Intake in Acute Decompensated Heart Failure
Acronym: RELIEF-AHF
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gødstrup Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1-16-02-56-26
Record Dates: First submitted 2026-02-03; First posted 2026-02-10 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Acute Heart Failure (AHF)
Keywords: Fluid Restriction; Thirst-driven fluid intake; Liberal fluid intake; Acute heart failure; Time to clinical stability

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Thirst-driven, liberal fluid intake (Experimental)
  Interventions: Behavioral: Thirst-driven, liberal fluid intake
- Fluid restriction (Active Comparator)
  Interventions: Behavioral: Fluid restriction strategy

INTERVENTIONS:
Behavioral: Fluid restriction strategy — Fluid restriction of 1.5 L/day
  Arms: Fluid restriction
Behavioral: Thirst-driven, liberal fluid intake — Liberal fluid intake driven by thirst without restrictions
  Arms: Thirst-driven, liberal fluid intake

SUMMARY:
The aim of this clinical trial is to learn whether a thirst-driven, liberal fluid-intake strategy is comparable to a fluid-restriction strategy in patients hospitalized for acute decompensated heart failure (ADHF). The study will also assess the safety of the intervention and its effects on thirst and quality of life.

Patients hospitalized with ADHF will be asked to follow either a thirst-driven fluid-intake strategy or a fluid-restriction strategy during their hospital stay and for one month after discharge.

ELIGIBILITY:
Inclusion Criteria:

1. Age >18 years
2. Hospitalized for ADHF as the primary diagnosis, meeting both of the following:

   1. ≥1 documented symptom of new or worsening heart failure (dyspnea, fatigue, decreased exercise tolerance, or symptom of end-organ hypoperfusion).
   2. Objective evidence of ADHF, defined as either:

   i. ≥2 physical signs (edema, ascites, pulmonary rales/crackles, increased JVP, S3 gallop, rapid weight gain due to fluid retention), OR ii. ≥1 physical sign AND ≥1 laboratory finding indicative of ADHF (BNP >500 ng/L or NT-proBNP >2000 ng/L if sinus rhythm, or BNP >750 ng/L or NT-proBNP >3000 ng/L if atrial fibrillation, radiological/ultrasound evidence of pulmonary congestion, echocardiographic sign [VCI >2.1 cm, LVOT VTI <15 cm, E/e' >14, D-dominant pulmonary venous inflow pattern], or invasive evidence [CVP >12 mmHg, PCWP >18 mmHg, CI <2.2 L/min/m2]).
3. Treatment with ≥40 mg IV furosemide (or equivalent)
4. Enrolment within 24 hours of admission
5. Ability to provide informed consent

Exclusion Criteria:

1. Requirement at admission for ICU-level care, or IV inotropic/vasopressor therapy for ADHF.
2. Na+ <125 mmol/L or Na+ >145 mmol/L.
3. End-stage chronic kidney disease on chronic dialysis or eGFR <15 mL/min/1.73 m2
4. Any condition which would make participation unsafe or substantially affect protocol adherence, as judged by investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Estimated)
Dates: Start 2026-05-01 (Estimated); Primary Completion 2029-05-01 (Estimated); Study Completion 2029-08 (Estimated)

PRIMARY OUTCOMES:
Time to clinical stability | From enrollment to 1 month follow-up
  Time from randomization to clinical stability. Clinical stability is defined as:
  1. Off IV loop diuretics for ≥ 24 hours without need for reinitiation of IV diuretics.
  2. No evidence of pulmonary congestion, defined as both:
     i) No new or worsening dyspnea at rest compared with status at admission ii) Clear lung auscultation or clinically improved, or normal lung and/or vena cava ultrasound without evidence of congestion.
  3. No new or worsening peripheral edema compared with status at admission.

SECONDARY OUTCOMES:
Thirst Distress | From enrollment to 1 month follow up
  Thirst Distress Scale for patients with Heart Failure (TDS-HF). Scores range from 8 to 40. Higher scores indicate greater thirst-related distress
Patient-perceived Quality of Life | From enrollment to 1 month follow up
  Kansas City Cardiomyopathy Questionnaire (KCCQ). Scores range from 0 to 100, with higher scores indicating better health status.
Incidence of Treatment-Emergent Adverse Events (Safety and Tolerability) | From enrollment to 1 month follow up
  Number of occurrences during hospitalization of clinical worsening (escalation of HF therapy, such as vasopressor/inotrope initiation, ICU transfer, dialysis, reinitiation of IV diuretics), electrolyte disturbances, worsening renal function, or in-hospital death, and similarly after one month including HF hospitalization

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Cardiology, Gødstrup Hospital, Herning, Denmark

IPD SHARING:
Plan to Share IPD: Undecided
Due to regulations by Region Committees on Health Research Ethics